CLINICAL TRIAL: NCT04863248
Title: A Phase 2 Randomized, Double-blind, Clinical Trial of Trilaciclib Versus Placebo in Patients With Metastatic Non-Small Cell Lung Cancer (NSCLC) Treated With Docetaxel in the 2nd/3rd Line Setting (PRESERVE 4)
Brief Title: Trilaciclib, a CDK 4/6 Inhibitor, in Patients Receiving Docetaxel for Metastatic Non-Small Cell Lung Cancer (NSCLC) (PRESERVE 4)
Acronym: PRESERVE 4
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Treatment paradigm in second- and third-line NSCLC is shifting away from docetaxel, the backbone chemotherapy therapy used in this study.
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G1T28-210; 2021-000186-32 (EudraCT Number)
Record Dates: First submitted 2021-04-16; First posted 2021-04-28 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Non-Small Cell Lung Cancer; NSCLC; Lung Cancer
Keywords: Trilaciclib; Lung Cancer; Non-Small Cell Lung Cancer; PRESERVE 4; CDK 4/6 Inhibitor; cyclin-dependent kinase 4/6 inhibitor; Preserve; NSCLC; solid tumors; chemotherapy; metastatic; myeloprotection; advanced; stage 4; lung; docetaxel; COSELA; G1T28
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis | interventions — trilaciclib; Sodium Chloride; Glucose; Water; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- trilaciclib + docetaxel (Experimental): Patients will receive trilaciclib administered IV prior to docetaxel administered IV on Day 1 of each 21-day cycle.
  Interventions: Drug: Trilaciclib; Drug: Docetaxel
- placebo + docetaxel (Placebo Comparator): Patients will receive placebo administered IV prior to docetaxel administered IV on Day 1 of each 21-day cycle.
  Interventions: Drug: Placebo; Drug: Docetaxel

INTERVENTIONS:
Drug: Trilaciclib — Trilaciclib administered IV over 30 minutes prior to docetaxel IV on Day 1 of each 21-day cycle.
  Other Names: COSELA; G1T28
  Arms: trilaciclib + docetaxel
Drug: Placebo — Placebo administered IV over 30 minutes prior to docetaxel IV on Day 1 of each 21-day cycle.
  Other Names: 0.9% sodium chloride; 5% Dextrose in water (D5W)
  Arms: placebo + docetaxel
Drug: Docetaxel — Docetaxel administered IV on Day 1 of each 21-day cycle.
  Other Names: Taxotere; Docefrez

SUMMARY:
This is a randomized, double-blind, placebo-controlled, global, multicenter, Phase 2 trial evaluating the effect of trilaciclib on overall survival when administered prior to docetaxel in patients with metastatic NSCLC treated in the 2nd or 3rd line setting.

DETAILED DESCRIPTION:
Patients must have documented disease progression during or after one or two lines of systemic therapy for recurrent or metastatic NSCLC. Prior treatment must have included, either in the same line or as separate lines of therapy: 1) a maximum of 1 line of platinum-containing chemotherapy for recurrent/metastatic disease and 2) a maximum of 1 line of a locally approved/authorized programmed cell death protein 1 (PD-1)/programmed death-ligand 1 (PD-L1) monoclonal antibody (mAb) containing regimen for recurrent/metastatic disease.

Patients will be randomly assigned (1:1) to receive trilaciclib or placebo intravenously (IV) prior to docetaxel on Day 1 of each 21-day cycle.

The study will include a screening phase, a treatment phase and a survival follow-up phase. The patient may continue to receive treatment on study until disease progression, unacceptable toxicity, withdrawal of consent, discontinuation by Investigator, or the end of the trial, whichever occurs first.

This study was terminated by the Sponsor for non-safety reasons. At the time of study termination, 10 patients had been screened, 7 were randomized, and 2 of the 7 had discontinued from the study. In addition, it was decided that there would be no statistical analyses of the efficacy or safety data due to the limited number of patients treated (N=7).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age at the time of signing the informed consent.
* Histologically or cytologically confirmed metastatic NSCLC (squamous or nonsquamous) with no known actionable driver mutations (eg, EGFR, ROS1, ALK).

  1. Patients must have had documented disease progression during or after 1 or 2 lines of systemic treatment for recurrent or metastatic disease.
  2. Two components of treatment must have been received in the same line or as separate lines of therapy: (i) a maximum of 1 line of platinum-containing chemotherapy regimen for recurrent/metastatic disease, and (ii) a maximum of 1 line of a locally approved/authorized PD-1/PD-L1 mAb containing regimen for recurrent/metastatic disease.
  3. Maintenance therapy following platinum doublet-based chemotherapy is not considered as a separate line of therapy. Maintenance therapy is defined as therapy given within 42 days after the last dose of platinum-based chemotherapy in patients with ongoing clinical benefit (complete response [CR], partial response [PR] or stable disease [SD]).
* Measurable or non-measurable disease per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
* A formalin-fixed paraffin-embedded (FFPE) tumor specimen (from archival or fresh biopsy) with an associated pathology report documenting NSCLC must be available to send to the Sponsor, within the specified timeframe, for planned retrospective biomarker analyses.
* Adequate organ function defined by the normal laboratory values.

Exclusion Criteria:

* Prior therapy with docetaxel.
* Any contraindication to the administration of docetaxel at the discretion of the investigator.
* Mixed NSCLC/SCLC, or lung tumors whose predominant histology is sarcomatoid, or neuroendocrine.
* Any chemotherapy, immunotherapy, biologic, investigational, or hormonal therapy for cancer treatment (except for adjuvant hormonal therapy for breast cancer or prostate cancer defined as M0 disease or prostate-specific antigen (PSA) persistence/recurrence without metastatic disease) within 3 weeks prior to the first dose of trilaciclib/placebo.
* Any radiotherapy within 2 weeks prior to the first dose of trilaciclib/placebo.
* Presence of central nervous system (CNS) metastases requiring immediate treatment with radiation therapy or steroids (i.e., patient must be off steroids administered for brain metastases for at least 14 days prior to the first dose of trilaciclib/placebo).
* Presence of leptomeningeal disease.
* Significant third-space fluid retention (eg, ascites or pleural effusion) not amenable to required repeat drainage.
* QT corrected using Fridericia's formula (QTcF) interval >480 msec at screening (confirmed on repeat). For patients with ventricular pacemakers, QTcF >500 msec.
* Symptomatic peripheral neuropathy.
* History of interstitial lung disease (ILD).
* Prior allogeneic or autologous hematopoietic stem cell or bone marrow transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Contact, Study Director — G1 Therapeutics, Inc.
Locations (12):
- United States (12):
  - Ironwood Cancer & Research Centers, Phoenix, Arizona
  - Valkyrie Clinical Trials, Los Angeles, California
  - Desert Hematology Oncology Medical Group, Inc, Rancho Mirage, California
  - Innovative Clinical Research Institute - Oncology, Whittier, California
  - Mid-Florida Hematology Oncology, Orange City, Florida
  - Indiana University Health Goshen Cancer Center, Goshen, Indiana
  - St. Louis Cancer Care, LLP, Bridgeton, Missouri
  - Summit Medical Group, Florham Park, New Jersey
  - Regional Cancer Car Associates, LLC, Little Silver, New Jersey
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Millennium Oncology, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to the rapidly evolving treatment landscape for patients with metastatic NSCLC, G1 Therapeutics announced the decision to terminate this study on 03 November 2021. This study was not terminated for reasons related to safety. At the time of study termination, 10 patients had been screened, 7 were randomized, and 2 of the 7 had already discontinued from the study.
Pre-assignment Details: Of the 10 patients enrolled, 3 were screen failures and 7 patients were randomized to treatment.
Groups:
- Trilaciclib + Docetaxel: Patients will receive trilaciclib administered IV no more than 4 hours prior to docetaxel administered IV on Day 1 of each 21-day cycle.
  Trilaciclib: Trilaciclib administered IV over 30 minutes prior to docetaxel IV on Day 1 of each 21-day cycle.
  Docetaxel: Docetaxel administered IV on Day 1 of each 21-day cycle.
- Placebo + Docetaxel: Patients will receive placebo administered IV no more than 4 hours prior to docetaxel administered IV on Day 1 of each 21-day cycle.
  Placebo: Placebo administered IV over 30 minutes prior to docetaxel IV on Day 1 of each 21-day cycle.
  Docetaxel: Docetaxel administered IV on Day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | Trilaciclib + Docetaxel | Placebo + Docetaxel
Started | 4 | 3
Completed | 0 | 0
Not Completed | 4 | 3
Not completed — Sponsor Terminated | 4 | 1
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trilaciclib + Docetaxel | Placebo + Docetaxel | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (11.47) | 62.7 (2.52) | 60.1 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG Score [Count of Participants; unit: Participants] — The ECOG Performance Status Scale describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.).
  Grade 0= Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1= Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Grade 2= Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    0 | 1 | 1 | 2
    1 | 2 | 2 | 4
    2 | 1 | 0 | 1
Stage at Diagnosis [Count of Participants; unit: Participants] — The stage at diagnosis measures how far the cancer has spread to other organs or parts of the body at the time it was detected.
  Stage IV: Metastatic; cancer has spread from where it originated in the lung to other parts of the body
  Participants
    IV | 4 | 3 | 7
    Unknown | 0 | 0 | 0
Histopathologic Type [Count of Participants; unit: Participants]
  Adenocarcinoma | 3 | 2 | 5
  Squamous Cell Carcinoma | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events as Assessed by CTCAE v5.0
Description: To assess the effects of trilaciclib administered prior to docetaxel compared with placebo administered prior to docetaxel on occurrence and severity of adverse events (AEs) by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5, study treatment discontinuation due to adverse events (AEs), and trilaciclib adverse events of special interest (AESI) in patients with metastatic NSCLC receiving docetaxel in the second or third line.
Time Frame: Time from date of first dose of trilaciclib/placebo and docetaxel through 30 days following the last dose of trilaciclib/placebo and docetaxel, assessed up to 9 months and 2 days.
Population: This study was terminated by the Sponsor for non-safety reasons. At the time of study termination, 10 patients had been screened, 7 were randomized, and 2 of the 7 had discontinued from the study. In addition, it was decided that there would be no statistical analyses of the efficacy or safety data due to the limited number of patients treated (N=7).
Measure: Number; unit: participants
Arm/Group | Trilaciclib + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 4 | 3
participants
  Any AE | 4 | 3
  Any AE of Grade >= 3 | 2 | 3
  Any AE of Grade >= 4 | 0 | 3

ADVERSE EVENTS:
Time Frame: 9 months, 2 days
Arm/Group | Trilaciclib + Docetaxel | Placebo + Docetaxel
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 3/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trilaciclib + Docetaxel (N=4) | Placebo + Docetaxel (N=3)
Staphylococcal sepsis (Infections and infestations) | 0 | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 | 1 (1)
Urosepsis (Infections and infestations) | 0 | 1 (1)
Renal failure (Renal and urinary disorders) | 0 | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trilaciclib + Docetaxel (N=4) | Placebo + Docetaxel (N=3)
Leukopenia (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Eosinopenia (Blood and lymphatic system disorders) | 1 | 2
Metamyelocyte count increased (Investigations) | 0 | 2
Monocytosis (Blood and lymphatic system disorders) | 2 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Neutrophilia (Blood and lymphatic system disorders) | 1 | 1
Protein total decreased (Investigations) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Monocytopenia (Blood and lymphatic system disorders) | 3 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Myelocyte count increased (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Cortisol increased (Investigations) | 0 | 1
Fatigue (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Early satiety (General disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Hyperchloremia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated earlier than initially proposed by the Sponsor for non-safety related reasons; only 7 patients were randomized and treated. Therefore, only limited safety summary tables were generated, and no efficacy analyses were conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT04863248/Prot_SAP_001.pdf